CLINICAL TRIAL: NCT04065607
Title: Professor and Head of Department of Surgery Dow University Hospital DUHS
Brief Title: Indications and Outcome of Laparostomy
Status: Completed | Type: Observational
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shahida Parveen Afridi, Professor and Head of Department of surgery, Dow University of Health Sciences
Other Study IDs: DIMC 233
Record Dates: First submitted 2019-08-10; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Laparotomy
Keywords: Laparotomy; Laparostomy; Open abdomen (OA); Temporary abdominal closure (TAC); Relook laparotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Reopen the abdomen to check missed pathology or abdominal washouts — Re opening of the abdomen once the patient is stabilized after 24-48 hours to check the missed injury after damaged control surgery in trauma and to control the sepsis in fecal peritonitis due to abdominal tuberculosis or typhoid perforation

SUMMARY:
Brief study Introduction/background Laparostomy is defined is a surgical procedure in which abdominal cavity is opened and left opened deliberately because of difficult primary closure or when primary closure is avoided due to severe intraabdominal sepsis, trauma and risk of abdominal compartment syndrome.

Patients and methods Retrospective Proforma based study conducted from 1st May 2014-31st May 2018. All patients admitted through emergency diagnosed clinically with peritonitis, intraabdominal sepsis and abdominal trauma managed with laparotomy and laparostomy were included in the study. On laparotomy primary cause was identified and controlled with damaged control surgery to save the lives and abdomen was left open with temporary abdominal wall cover of urine bag stitched all around either with skin or external oblique aponeurosis temporarily for second relook laparotomy after 24-48 hours. On second relook of abdomen haemostasis secured and abdomen was washed with normal saline, any missed pathology identified and controlled and abdomen was closed in some patient when there was no need to recheck the abdomen while in other patients abdominal content were covered again temporarily with urine bag. All patients were managed by the team of surgery and ICU. Finally abdomen was closed by deep tension suture DTS or direct layered closure of abdominal wall.

DETAILED DESCRIPTION:
Detail study Introduction Laparostomy is a surgical procedure in which abdominal cavity is opened and left opened deliberately called open abdomen, an open abdomen is based on the principle of incision and drainage of an abscess and leaving the wound open for free drainage, washouts and multiple dressings1.

Usually abdomen is closed primarily in all abdominal surgeries but some time it is difficult to close the abdomen primarily to avoid intraabdominal hypertension because the risk of abdominal compartment syndrome and to manage severe intraabdominal sepsis2. Trauma required damage control surgery 3, and other complex abdominal pathologies, injuries due to explosive devices4, laparostomy and finally staged abdominal closure or DTS deep tension sutures are used to close the abdomen5. Multiple techniques are used to close the abdomen temporarily after laparotomy to have a second relook laparotomy6. Laparostomy is a complex procedure and it is difficult to identify which is the best technique for temporary abdominal closure, primary fascial closure, mesh, plastic sheet, bagota bag, urine bag, vacuum assisted closure are commonly used methods to cover the abdominal content to prevent the risk of injury evisceration and direct exposure to the atmosphere7.

Our objective is to identify the indications and outcome of laparostomy in emergency laparotomy and prevent the abdominal compartment syndrome, in critically ill patients due to fecal peritonitis, intraabdominal sepsis and trauma.

Patients and methods Retrospective Proforma based study conducted from 1st May 2014-31st May 2018 at Dow International Hospital Ojha Campus Dow University of Health Sciences Karachi Pakistan.

Inclusion Criteria: all critically ill patients admitted through emergency, diagnosed with peritonitis, intraabdominal sepsis and trauma managed with damaged control surgery initially along with laparostomy in which the abdomen was left open with temporary abdominal cover to have a relook laparotomy were included in the study Exclusion Criteria: Patients diagnosed clinically with peritonitis and trauma but managed by primary abdominal wall closure were excluded from the study.

Initially all Patients were optimized and resuscitated and all necessary investigations were send in emergency eg blood grouping and cross matching, blood complete picture, serum electrolyte ,blood urea & creatinine screening for hepatitis. Antibiotic cover, fluid and electrolyte support was given to all patients. FFP arranged according to the requirement. Imaging performed where necessary in stable patients.

On laparotomy primary cause was identified and managed with damaged control surgery along with abdominal washout and abdomen was covered with a urine bag open from the center to make a sheet then sutured all around with the skin or external oblique aponeurosis. All patients were managed in the ICU initially for a second relook laparotomy.

Second relook laparotomy was performed after 24-48 hours abdomen was washed with normal saline haemostasis secured and any missed primary pathology was identified and controlled. Abdomen was closed in few patient where no need to recheck the abdomen, while in remaining patients abdominal content were covered again with urine bag who require multiple washouts and dressing. All patients managed by the team of ICU, anesthesia, surgeon, and physician from critical care medicine. Morbidity and mortality happen recorded during the period of hospital stay Patient discharged after complete recovery with the final closure of abdominal wall either with deep tension suture DTS figure 4 or direct layered closure of abdominal wall. Data was collected and recorded on a pre designed research Proforma made for this study. SPSS version 20 was used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted through emergency surgery, diagnosed with fecal peritonitis
* Intraabdominal sepsis due to tuberculosis & typhoid perforation
* Trauma managed with damaged control surgery need a relook laparotomy

Exclusion Criteria:

* Patients diagnosed clinically with peritonitis and traumas, managed by primary abdominal wall closure were excluded from the study.
* Age below 20 years
* Age above 70 years

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ll Emergency surgery and intensive care admission who require exploratory laparotomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Indications of Laparostomy | Duration of study: 1st May 2014-31st May 2018.
  Conditions or disease for which laparostomy performed
Mortality | Two months
  Mortality happen during hospital stay

SECONDARY OUTCOMES:
Chest infection | Two months
  Chest infection during the admission in hospital
Abdominal wall surgical site infection | Four months
  Infection of abdominal wall during hospital admission or after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Shahida Afridi, FCPS, Principal Investigator — HOD of Surgery Dow University Hospital .Dow University of Health Sciences; Naveed Khan, FCPS,MRCS, Study Chair — Assciate Professor Surgery Dow University of Health Sciences

IPD SHARING:
Plan to Share IPD: Yes
Study can be shared after the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One month after the publication
Access Criteria: pubmed id